CLINICAL TRIAL: NCT05291741
Title: Use of Very Low Calorie Diet Preoperatively to Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-16-02-436-21
Record Dates: First submitted 2022-02-21; First posted 2022-03-23 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Bariatric Surgery Candidate; Very Low Calorie Diet; Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Very Low Calorie Diet (VLCD) (Active Comparator): VLCD
  Interventions: Dietary Supplement: VLCD
- Standard care (Placebo Comparator): Standard care
  Interventions: Dietary Supplement: Standard care

INTERVENTIONS:
Dietary Supplement: VLCD — Advice regarding VLCD
  Arms: Very Low Calorie Diet (VLCD)
Dietary Supplement: Standard care — Standard dietary advice for weight loss before bariatric surgery
  Arms: Standard care

SUMMARY:
To investigate use of Very Low Calorie Diet preoperatively to bariatric surgery can optimize weight loss prior to surgery and increase the patients' satisfaction.

DETAILED DESCRIPTION:
In this project the investigators want to develop an effective Very Low Calorie Diet (VLCD) treatment prior to bariatric surgery, which is optimized in relation to the size and speed of the weight loss as well as in terms of satisfaction both for the patients as for the health care professionals. Thus the investigators will randomize 500 patients to either VLCD or standard care prior to bariatric surgery. The investigators aim to optimize preoperative and the operative course for patients, who are offered bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for bariatric surgery

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 8 weeks

SECONDARY OUTCOMES:
Patient quality of life measured using the Short Form-12 (SF-12) questionnaire | 8 weeks and 1 year
  Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Positive and negative consequences of the two weight loss treatments identified by the surgeon, using a questionnaire developed for the purpose | 30 days after surgery
  In the questionnaire, the surgeon will be asked questions on details on the surgery, including duration of surgery and complicating factors.
Use of health care services assessed by a medical chart review | 30 days after surgery
  We will assess the number of health care contacts for each patient.
Severity of complications assessed by a medical chart review. | 30 days after surgery
  We will define the severity of the contacts based on whether they are outpatient or inpatient contacts.
Presence of eating disorders | At baseline
  The patients will be asked to complete the Eating Disorder Examination Questionnaire (EDE-Q) to assess whether diorderes eating is present. Scores range from 0 to 6 and a score of 4 and above indicate disordered eating.

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No